CLINICAL TRIAL: NCT02360059
Title: Metformin for Reduction of Paclitaxel Treatment-Related Neuropathy in Patients With Breast Cancer: A Randomized Pilot Study
Brief Title: Metformin for Reduction of Paclitaxel-Related Neuropathy in Patients With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-0438; NCI-2015-00510 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Neuropathy; Paclitaxel; Metformin; Metformin ER; Placebo; Sugar pill; Questionnaires; Sensory tests; Fine-motor tests; Surveys
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin; Sugars; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin Group (Experimental): Participants take 1,000 mg Metformin by mouth twice daily for 12 weeks during Paclitaxel treatment.
  Adaptation phase begins 12 days prior to the start of the Paclitaxel therapy. During this phase, study medication dose starts at 500 mg daily for 5 days, followed by 500 mg twice daily for 5 days, followed by the desired dose of 1,000 mg twice daily for 2 days. Participants reach required study medication dose of 2,000 mg daily 2 days prior to commencement of Paclitaxel therapy and continue this dose for remainder of intervention.
  Questionnaires completed about numbness and/or symptoms about 2 weeks before start of Paclitaxel, 1 -2 days before Paclitaxel, every week while taking Paclitaxel, and at end of study visit. At week 12, questionnaire completed regarding satisfaction with Paclitaxel.
  Three sensory and fine-motor tests completed 2 weeks before Paclitaxel, every 3 weeks while taking Paclitaxel, and at end of study visit.
  Interventions: Drug: Metformin; Behavioral: Questionnaires; Other: Sensory and Fine-Motor Tests
- Placebo Group (Placebo Comparator): Participants take placebo by mouth twice daily starting 12 days before, and 12 weeks during Paclitaxel treatment.
  Questionnaires completed about numbness and/or symptoms about 2 weeks before start of Paclitaxel, 1 -2 days before Paclitaxel, every week while taking Paclitaxel, and at end of study visit. At week 12, questionnaire completed regarding satisfaction with Paclitaxel.
  Three sensory and fine-motor tests completed 2 weeks before Paclitaxel, every 3 weeks while taking Paclitaxel, and at end of study visit.
  Interventions: Other: Placebo; Behavioral: Questionnaires; Other: Sensory and Fine-Motor Tests

INTERVENTIONS:
Drug: Metformin — Metformin dose starts at 500 mg daily for 5 days, followed by 500 mg twice daily for 5 days, followed by 1,000 mg twice daily for 2 days. Participants reach required study medication dose of 2,000 mg daily 2 days prior to commencement of Paclitaxel therapy and continue this dose for remainder of intervention.
  Other Names: Metformin ER
  Arms: Metformin Group
Other: Placebo — Participants take placebo by mouth twice daily starting 12 days before, and 12 weeks during Paclitaxel treatment.
  Other Names: Sugar pill
  Arms: Placebo Group
Behavioral: Questionnaires — Questionnaires completed about numbness and/or symptoms about 2 weeks before start of Paclitaxel, 1 -2 days before Paclitaxel, every week while taking Paclitaxel, and at end of study visit. At week 12, questionnaire completed regarding satisfaction with Paclitaxel.
  Other Names: Surveys
Other: Sensory and Fine-Motor Tests — Three sensory and fine-motor tests completed 2 weeks before Paclitaxel, every 3 weeks while taking Paclitaxel, and at end of study visit.

SUMMARY:
The goal of this clinical research study is to learn if metformin can help to control nerve damage (loss of motor or sensory function) that may be caused by treatment with paclitaxel in patients with breast cancer.

In this study, metformin will be compared to a placebo. A placebo is not a drug. It looks like the study drug, but it is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in a roll of dice) to 1 of 2 groups. This is done because no one knows if one study group is better, the same, or worse than the other group. You will have a 1 out of 3 chance of being in Group 1 and a 2 out of 3 chance of being in Group 2.

* If you are in Group 1, you will take placebo pills.
* If you are in Group 2, you will take metformin pills.

Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Drug Administration:

You should take the pills 2 times a day at about the same time every day, preferably with food (for example, with breakfast and dinner).

You will start taking the pills about 12 days before your paclitaxel treatment starts. This is called the "adaptation period." It is meant to allow your body to get used to the study pills. The study staff will check you for allergic reactions or other negative reactions to the pills during this period. If you are not tolerating the pills, you will be taken off study.

About every 3 weeks while you are receiving paclitaxel, you should bring the study drug/placebo container (along with any leftover pills) to the clinic. The study staff will count the number of pills you have taken.

Study Visits:

Every week during the study, either during your clinic visit or by phone, the study staff will ask you about any side effects you may be having, if you have taken the study drug/placebo, and how many pills you have taken so far. The calls should take about 10-15 minutes.

About 2 weeks before you start paclitaxel:

* You will complete questionnaires about numbness and other symptoms. It should take about 15 minutes to complete these questionnaires.
* You will complete 3 sensory and fine-motor tests. These tests will show researchers how sensitive you are to touching things such as small bumps and how well you are able to pick up small objects. It should take about 15 minutes to complete these tests.
* If possible, blood (about 8 teaspoons) will also be drawn to test for markers of inflammation. Markers of inflammation are biomarkers found in the blood and may be related to the symptoms you have. These blood samples during the study will only be collected if they can be drawn during a routine blood draw you are already having.

At 1-2 days before you start paclitaxel:

* You will complete the questionnaires about numbness and other symptoms.
* You will complete the sensory and fine-motor tests.
* Blood (about 8 teaspoons) will be drawn to test for markers of inflammation, if a routine blood sample is also being drawn on that day.

Every week while you are receiving paclitaxel, you will complete a questionnaire in the clinic or by phone about any symptoms you may be having, and how the symptoms may be affecting your daily activities. This questionnaire should take about 5 minutes to complete.

About every 3 weeks while you are receiving paclitaxel, at your clinic visits:

* You will complete the questionnaires about numbness.
* You will also complete the sensory and fine-motor dexterity tests.

At about Weeks 6 and 12 while you are receiving paclitaxel, at your clinic visits, blood (about 8 teaspoons) will be drawn to test for markers of inflammation, if a routine blood sample is also being drawn on that day.

At about Week 12 while you are receiving paclitaxel, at your clinic visit, you will complete a questionnaire about how satisfied you are with the study drug/placebo. Completing the questionnaire should take about 5 minutes.

Length of Study:

You may take the study drug/placebo for up to 12 weeks. You will no longer be able to take the study drug/placebo if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation in the study will be over after the end-of-study visit.

End-of-Study Visit:

About 4 weeks after you finish receiving the study drug/placebo:

* You will complete the questionnaires about numbness and other symptoms.
* You will complete the sensory and fine-motor tests.
* Blood (about 8 teaspoons) will be drawn to test for markers of inflammation, if a routine blood sample is also being drawn on that day.

This is an investigational study. Metformin is FDA approved and commercially available for the treatment of a type of diabetes. Its use in this study is investigational. The study doctor can explain how the study drug is designed to work.

Up to 42 participants will be enrolled in this study. All will take part at the Harris Health System.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed invasive breast cancer, stage I - IV, treated at Lyndon B. Johnson General Hospital in the Harris Health System.
2. Patients = or > 18 years old and < 75 years old.
3. Patients scheduled to undergo paclitaxel chemotherapy for breast cancer.
4. Patients with adequate renal function, as evidenced in laboratory values = or < 3 months old: epidermal growth factor receptor (eGFR) = or > 60 mL/min/1.73m2.
5. Patients with adequate hepatic function per institutional testing standards, as evidenced in laboratory values = or < 3 months old: (1) The screening results for total bilirubin must be < 1.5 times the upper limit of normal. (2) The screening results for aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be < 2 times the upper limit of normal.
6. Patients who speak English and/or Spanish.
7. Patients who are willing and able to review, understand, and provide written consent.
8. Patients with an Eastern Cooperative Oncology performance status of 0 or 1.

Exclusion Criteria:

1. Patients with a history of or known diagnosis of diabetes according to national guidelines (fasting plasma glucose > or = 126 mg/dL or random plasma glucose > or = 200 mg/dL), as evidenced in laboratory values < or = 3 months old).
2. Patients using carbonic anhydrase inhibitors (acetazolamide [Diamox®], brinzolamide [Azopt®], methazolamide [Neptazane®], dorzolamide [Trusopt®], pomegranate ellagitannins), cimetidine, or topiramate.
3. Patients who are enrolled in another symptom management trial.
4. Patients with nerve pathology or clinically identified neuropathy.
5. Patients with a history of clinically significant cutaneous drug reaction, hypersensitivity reaction, anaphylaxis, or any other serious adverse reaction to the medication used in the study.
6. Patients with any condition associated with increased risk of metformin-associated lactic acidosis (e.g., congestive heart failure defined as New York Heart Association Class III or IV functional status, history of acidosis of any type).
7. Patients with intestinal issues, including malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel.
8. Patients who are pregnant are excluded. Pre-menopausal women must have a negative pregnancy test. Patients that are post menopausal, or that have had a hysterectomy do not need to have a pregnancy test.
9. Patients with any condition that precludes use of the study medication as determined by the treating physician.
10. Patients with a diagnosis of hepatitis or HIV.
11. Patients currently receiving or scheduled to receive a chemotherapy infusion other than Adriamycin/Cyclophosphamide prior to initiation of the metformin adaptation phase are not eligible. Patients who are receiving Adriamycin/Cyclophosphamide must be scheduled to be at least 8 days post-chemotherapy infusion prior to initiation of the metformin adaptation phase in order to be eligible.
12. Patients who are currently using metformin (eg, Fortamet, Glucophage, Glucophage XR, Glumetza, Riomet).

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L. Ramirez, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Lyndon B. Johnson General Hospital, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 06, 2015 to July 22, 2016. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Changes in breast cancer treatment and this study's requirement for a long rest-interval led to lower than expected accrual rate resulting in early study termination.
Groups:
- Metformin Group: Participants take 1,000 mg Metformin by mouth twice daily for 12 weeks during Paclitaxel treatment.
- Placebo Group: Participants take placebo by mouth twice daily starting 12 days before, and 12 weeks during Paclitaxel treatment.
Period: Overall Study
Arm/Group | Metformin Group | Placebo Group
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin Group | Placebo Group | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Neuropathy
Description: Change in neuropathy as assessed with the chemotherapy-induced peripheral neuropathy (CIPN) survey QLQ-CIPN20 between T1 and T5 where difference in mean area under the curve (AUC) between groups reported. The AUC for response from T1 to T5 is computed by fitting a series of trapezoids to the QLQ-CIPN20 data assessed at T1, T2, T3, T4, and T5, respectively, and summing up their areas [AUC calculated - base of a trapezoid corresponds to the number of days between assessments, and the heights correspond to two adjoining symptom responses, number of trapezoids depends on number of symptom assessments and sum of area for all trapezoids represents AUC of particular participant]. QLQ-CIPN20 contains 20 items assessing sensory (9 items), motor (8 items), and autonomic symptoms (3 items) using a 4-point Likert scale (1 = "not at all," 2 = "a little," 3 = "quite a bit," and 4 = "very much") with the higher score denoting more symptom burden.
Time Frame: Up to 14 weeks, assessed every 3 weeks ±1 week (T2, T3, T4, T5) during paclitaxel therapy
Population: Study stopped early with only one participant, analysis not possible.
Arm/Group | Metformin Group | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collected was up to 18.5 weeks (13.5 weeks of intervention and 4 ± 1week after end of treatment).
Arm/Group | Metformin Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes